CLINICAL TRIAL: NCT02063529
Title: A Phase II Study to Evaluate the Surgical Conversion Rate in Patients Receiving FOLFOXIRI +/- Cetuximab for Unresectable Wild-Type KRAS/NRAS Colorectal Cancer With Metastases Confined to the Liver
Brief Title: FOLFOXIRI With or Without Cetuximab as First-line Treatment of Patients With Non-resectable Liver - Only Metastatic Colorectal Cancer
Acronym: FOCULM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Associate professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU05
Record Dates: First submitted 2014-02-08; First posted 2014-02-14 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Metastatic colorectal cancer; Liver metastases; Liver resection; Liver ablation; Conversion therapy; FOLFOXIRI; Cetuximab; Oxaliplatin; Irinotecan; Leucovorin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil; FOLFOXIRI protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (FOLFOXIRI + Cetuximab) (Experimental): FOLFOXIRI + Cetuximab
  Interventions: Drug: FOLFOXIRI + Cetuximab
- B (FOLFOXIRI) (Active Comparator): FOLFOXIRI
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI + Cetuximab — Cetuximab 500mg/m² + irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle until PD or resectability or to max. 12 cycles
  Other Names: Cetuximab; Irinotecan; Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: A (FOLFOXIRI + Cetuximab)
Drug: FOLFOXIRI — Irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle until PD or resectability or to max. 12 cycles
  Other Names: Irinotecan; Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: B (FOLFOXIRI)

SUMMARY:
PURPOSE:

A primary aim of phase II FOCULM study is to explore whether cetuximab in combination with FOLFOXIRI as first treatment could improve surgical conversion in patients with KRAS/NRAS wild-type, unresectable liver - only metastases of colorectal cancer. The first secondary aim is to evaluate the safety and tolerability of the chemotherapy of FOLFOXIRI plus Cetuximab targeted therapy regimen in this patient population.

Secondary aims include determination of objective response rate, progression free survival, quality of life and time to recurrence for patients undergoing complete resection and/or ablation of liver.

DETAILED DESCRIPTION:
Patients will be randomized to two therapy groups:

Experimental arm A: Chemotherapy with FOLFOXIRI + Cetuximab Standard arm B: Chemotherapy with FOLFOXIRI

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study specific procedures. Subjects must be able to understand and willing to sign a written informed consent.
* Male or female subjects > 18 years < 65 of age
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and must be considered a potential candidate for a major hepatic surgical procedure.
* Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
* There must be documentation by PET/CT scan, CT scan, MRI, or intraoperative palpation (at the time of resection of the primary colorectal tumor, if applicable) that the patient has evidence of metastases confined to the Liver (Histologic confirmation of hepatic metastasis is not required.). The liver metastases must have been determined by a hepatic surgeon approved to participate in the study to be unresectable based on at least one of the following criteria: All of the liver metastases can not be resected (and/or ablated) with negative margins, i.e., lesion(s) located in an area that would result in the resection of all of the hepatic veins or the main portal vein or the right and left hepatic arteries or the common bile duct; Complete resection and/or ablation would require greater than 60% of the liver parenchyma to be removed.
* Patients are eligible with any of the following: primary tumor and regional nodes resected with clear surgical margins and no evidence of extra-hepatic disease or; unresected primary tumor with plans to resect the primary tumor prior to study entry or; unresected primary tumor with plans to resect the primary tumor and the liver metastases in a single surgical procedure performed within 8 weeks after the last preoperative dose of chemotherapy/cetuximab or; unresected primary with plans to resect the primary tumor and the liver metastases in staged procedures performed within 8 weeks after the last preoperative dose of chemotherapy/cetuximab.
* The colorectal primary tumor or metastatic tumor must be determined to be KRAS and NRAS wild-type.
* At least one measurable lesion in liver metastases according to according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria measured within 4 weeks prior to registration.
* No previous any systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy and hormonal therapy for metastatic disease for metastatic disease (adjuvant chemotherapy for non-metastatic disease is allowed if terminated more than 6 months ago).
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:
* Leukocytes ≥ 3.0 x109/ L, absolute neutrophil count (ANC) ≥ 1.5 x109/ L, platelet count ≥ 100 x109/ L, hemoglobin (Hb) ≥ 9g/ dL.
* Total bilirubin ≤1.5 x the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
* Alkaline phosphatase limit ≤ 5x ULN.
* Amylase and lipase ≤ 1.5 x the ULN.
* Serum creatinine ≤ 1.5 x the ULN.
* Calculated creatinine clearance or 24 hour creatinine clearance ≥ 50 mL/ min.

Exclusion Criteria:

* Any evidence of extra-hepatic metastases, lymph node (including portal lymph nodes) metastases and primary tumor recurrence.
* Previous hepatic resection and/or ablation, hepatic arterial infusion therapy, radiation therapy to the liver (Patients who have only had an excisional biopsy are eligible).
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization.
* Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to randomization. Subjects must have recovered from all therapy-related toxicities.
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks before start of study medication.
* Uncontrolled hypertension. (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment or a history of ventricular arrhythmia
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication.
* Any evidence of active infection.
* Known history of human immunodeficiency virus (HIV) infection.
* Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
* History of bleeding diathesis or coagulopathy.
* Uncontrolled hypertension. (systolic blood pressure ﹥150 mmHg or diastolic pressure ﹥ 90 mmHg despite optimal medical management).
* History of interstitial pneumonitis or pulmonary fibrosis
* Pregnancy or lactation at the time of study entry.
* Any history of or currently known brain metastases.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Any illness or medical conditions that are unstable or could jeopardize the safety of the subjects and his/her compliance in the study.
* Unresolved toxicity higher than CTCAE v. 4.0 Grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neurotoxicity ﹥ Grade 2.
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea
* Subjects with known allergy to the study drugs or to any of its excipients.
* Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-02; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
the percentage of patients who had a curative liver treatment following protocol treatment, i.e., liver metastases that can be completely resected and/or ablated with no evidence of residual malignant disease. | 8 months

SECONDARY OUTCOMES:
Reported adverse events. | 8 months
  Number of patients with adverse events and severity according to NCI CTC 4.0
Response rate | 8 months
  CR + PR rate according to RECIST
Progression free survival | 2 years
  Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first.
Time to recurrence | 2 years
  Time from date of complete resection and/or ablation of liver until first recurrence
Quality of life (QLQ C30) | Every 2 weeks after the first treatment until 6 months
  scores according to EORTC QLQ-C30 scoring manual

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China